CLINICAL TRIAL: NCT04184180
Title: Effects of an Inpatient Pulmonary Rehabilitation Programme on Frailty in Patients After Lung-Transplantation
Brief Title: Effects of Inpatient Pulmonary Rehabilitation on Frailty in Patients After Lung-Transplantation
Status: Completed | Type: Observational
Sponsor: Klaus Kenn (Other)
Responsible Party: Sponsor-Investigator, Klaus Kenn, Professor of pulmonary rehabilitation, Schön Klinik Berchtesgadener Land
Organization: Schön Klinik Berchtesgadener Land (Other)
Other Study IDs: Frailty post-LTx
Record Dates: First submitted 2019-10-23; First posted 2019-12-03 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-11

CONDITIONS: Advanced Lung Disease; COPD; Interstitial Lung Disease
Keywords: lung transplantation; pulmonary rehabilitation; exercise training; frailty; lung diseases; respiratory tract diseases
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases, Interstitial; Frailty; Lung Diseases; Respiratory Tract Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Frailty is closely linked to the success of lung transplantations (LTx) (1,2). Studies have shown that frailty causes a diminished physical performance in candidates for LTx and an increased 30 day rate of re-hospitalization after surgery. Furthermore, frailty is associated with a higher one-year-mortality rate after LTx in frail compared to non-frail patients (1,3,4).

Some evidence that frailty in LTx-candidates can be decreased by a suitable rehabilitation program suggests that improving the frailty status in post-LTx patients can be a further strategy to contribute to an overall success in LTx. However, at the moment these possible benefits are not investigated yet. Therefore the aim of this study is to observe the effect of a three-week inpatient rehabilitation on frailty in patients after LTx.

DETAILED DESCRIPTION:
Rationale:

Frailty is a complex clinical syndrome describing a loss of physical and/or cognitive functionality which leads to a decreased resistance to stressors such as operations or illness. It is associated with increased number of falls, exacerbations, adverse health outcomes and a higher mortality (7-10).

Frail LTx-candidates have a higher risk of being delisted before transplantation, adverse transplantation outcomes and a higher one-year-mortality compared to non-frail candidates. However, studies show that frailty can be decreased by physical training (11-13). A recent prospective cohort study in the UK observed a significant decrease of frailty in patients with COPD participating at an inpatient rehabilitation program (5). Singer et al. (USA) could detect a significant decrease of frailty by a homebased training for LTx-candidates (6).

Aim of this study is to investigate the effects of a three-week inpatient rehabilitation program on physical frailty (measured by Short Physical Performance Battery) in patients after LTx. Additionally, other functional measures as well as the cognitive, social and psychological state will be assessed in order to better understand the complex syndrome of frailty and the effects of rehabilitation.

Design:

This study is a prospective observational trial. The number of 30 participants is based on a sample size calculation. Assessments will take place in the beginning of rehabilitation program and at discharge.

ELIGIBILITY:
Inclusion Criteria:

* Participation in an inpatient pulmonary rehabilitation programme (Schön Klinik BGL, Germany)
* Patient after Lung Transplant (< 1 year)
* Indication: COPD or ILD
* written informed consent

Exclusion Criteria:

* Non compliance at assessments
* Re-Transplantation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be recruited during an inpatient pulmonary rehabilitation programme
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2019-12-02 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2020-03-16 (Actual)

PRIMARY OUTCOMES:
Change of Frailty (SPPB) | Day 1 and Day 21
  measured by Short Physical Performance Battery (SPPB) including three measurements (Balance, Gait Speed, Chair-Rising-Test); range 0-12, lower scores reflect increased Frailty

SECONDARY OUTCOMES:
Change of Frailty (FFP) | Day 1 and Day 21
  measured by Fried Frailty Phenotype (FFP), including five constructs (weight loss, exhaustion, physical activity, gait speed and weakness); range 0-5, higher scores reflect increased Frailty
Effect of Frailty on Six-Minute-Walking-Test (6MWT) | Day 1 and Day 21
  Frailty measured by Short physical Performance battery (SPPB)
Effect of Frailty on Timed-Up-an-Go-Test | Day 1 and Day 21
  Frailty measured by Short physical Performance battery (SPPB)
Effect of Frailty on Quadriceps-Force | Day 1 and Day 21
  Frailty measured by SPPB
Correlation between Frailty-Score (measured by Short physical Performance Battery (SPPB)) and attended exerecise sessions | Day 1 to Day 21
  Frailty socre will be measured by the Short physical Performance battery (SPPB); attended exercise sessions (number) will be assessed within the pulmonary Rehabilitation Programme.
Correlation between Cognitive Status measured by Montreal Cognitive Assessment (MOCA) and Frailty Score | Day 1
  Screening test for detecting cognitive impairment: including testing of orientation, memory, attention, language, visuospatial and executive skills and skills of abstraction; score 0-30; higher scores indicating better cognitive functioning; a score higher than 25 is considered as "normal"
Correlation between Cognitive Status measured by Addenbrooke's Cognitive Examination (ACE-R) and Frailty Score | Day 1
  the test allows more detailed information about the test person's cognitive functioning: including testing of attention, memory, verbal fluency, language and visuospatial abilities; score 0-100; higher scores indicating better cognitive functioning; a score higher than 86 is considered as "normal"
Correlation between Social Support and Frailty Score | Day 1 and Day 21
  Social Support measured by Oslo-3-Items-Social-Support Scale (Oslo-3); a 3-item self-report questionnaire ranging 3-14; higher scores reflecting higher social support
Change of Health related Quality of Life: Chronic Respiratory Questionnaire (CRQ) | Day 1 and Day 21
  measured by Chronic Respiratory Questionnaire (CRQ) - a 20-item self-report questionnaire; score 1-7; higher scores indicate a better health-related quality of life
Change of Fatigue | Day 1 and Day 21
  measured bei Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) - a self-report questionnaire including 40 items and ranging 0-160; higher scores indicating a higher Quality of life
Change of Anxiety/Depression | Day 1 and Day 21
  Anxiety/Depression measured by Hospital Anxiety and Depression Scale (HADS) - a screening questionnaire including seven questions each about Depression and Anxiety; each part ranging from 0 to 21; higher scores indicate higher presence of the respective state
Change of Sleeping Quality: Pittsburgh Sleep Quality Index (PSQI) | Day 1 and Day 21
  measured by Pittsburgh Sleep Quality Index (PSQI) - self-report questionnaire including seven components; score 0-21; lower scores indicating better sleep quality

CONTACTS AND LOCATIONS:
Locations (1):
- Schön Klinik Berchtesgadener Land, Schönau am Königssee, Germany

REFERENCES:
- [Background] Singer JP, Diamond JM, Gries CJ, McDonnough J, Blanc PD, Shah R, Dean MY, Hersh B, Wolters PJ, Tokman S, Arcasoy SM, Ramphal K, Greenland JR, Smith N, Heffernan P, Shah L, Shrestha P, Golden JA, Blumenthal NP, Huang D, Sonett J, Hays S, Oyster M, Katz PP, Robbins H, Brown M, Leard LE, Kukreja J, Bacchetta M, Bush E, D'Ovidio F, Rushefski M, Raza K, Christie JD, Lederer DJ. Frailty Phenotypes, Disability, and Outcomes in Adult Candidates for Lung Transplantation. Am J Respir Crit Care Med. 2015 Dec 1;192(11):1325-34. doi: 10.1164/rccm.201506-1150OC. PMID 26258797
- [Background] Milne KM, Kwan JM, Guler S, Winstone TA, Le A, Khalil N, Camp PG, Wilcox PG, Ryerson CJ. Frailty is common and strongly associated with dyspnoea severity in fibrotic interstitial lung disease. Respirology. 2017 May;22(4):728-734. doi: 10.1111/resp.12944. Epub 2016 Nov 9. PMID 27860036
- [Background] Singer JP, Diamond JM, Anderson MR, Katz PP, Covinsky K, Oyster M, Blue T, Soong A, Kalman L, Shrestha P, Arcasoy SM, Greenland JR, Shah L, Kukreja J, Blumenthal NP, Easthausen I, Golden JA, McBurnie A, Cantu E, Sonett J, Hays S, Robbins H, Raza K, Bacchetta M, Shah RJ, D'Ovidio F, Venado A, Christie JD, Lederer DJ. Frailty phenotypes and mortality after lung transplantation: A prospective cohort study. Am J Transplant. 2018 Aug;18(8):1995-2004. doi: 10.1111/ajt.14873. Epub 2018 May 14. PMID 29667786
- [Background] Courtwright AM, Zaleski D, Gardo L, Ahya VN, Christie JD, Crespo M, Hadjiliadis D, Lee J, Molina M, Patel N, Porteous M, Cantu EE, Bermudez C, Diamond JM. Causes, Preventability, and Cost of Unplanned Rehospitalizations Within 30 Days of Discharge After Lung Transplantation. Transplantation. 2018 May;102(5):838-844. doi: 10.1097/TP.0000000000002101. PMID 29346256
- [Background] Maddocks M, Kon SS, Canavan JL, Jones SE, Nolan CM, Labey A, Polkey MI, Man WD. Physical frailty and pulmonary rehabilitation in COPD: a prospective cohort study. Thorax. 2016 Nov;71(11):988-995. doi: 10.1136/thoraxjnl-2016-208460. Epub 2016 Jun 12. PMID 27293209
- [Background] Singer JP, Soong A, Bruun A, Bracha A, Chin G, Hays SR, Kukreja J, Rigler J, Golden JA, Greenland JR, Garvey C. A mobile health technology enabled home-based intervention to treat frailty in adult lung transplant candidates: A pilot study. Clin Transplant. 2018 Jun;32(6):e13274. doi: 10.1111/ctr.13274. Epub 2018 Jun 20. PMID 29742287
- [Background] Makary MA, Segev DL, Pronovost PJ, Syin D, Bandeen-Roche K, Patel P, Takenaga R, Devgan L, Holzmueller CG, Tian J, Fried LP. Frailty as a predictor of surgical outcomes in older patients. J Am Coll Surg. 2010 Jun;210(6):901-8. doi: 10.1016/j.jamcollsurg.2010.01.028. Epub 2010 Apr 28. PMID 20510798
- [Background] Rockwood K, Song X, Mitnitski A. Changes in relative fitness and frailty across the adult lifespan: evidence from the Canadian National Population Health Survey. CMAJ. 2011 May 17;183(8):E487-94. doi: 10.1503/cmaj.101271. Epub 2011 Apr 26. PMID 21540166
- [Background] Speechley M, Tinetti M. Falls and injuries in frail and vigorous community elderly persons. J Am Geriatr Soc. 1991 Jan;39(1):46-52. doi: 10.1111/j.1532-5415.1991.tb05905.x. PMID 1987256
- [Background] McIsaac DI, Taljaard M, Bryson GL, Beaule PE, Gagne S, Hamilton G, Hladkowicz E, Huang A, Joanisse JA, Lavallee LT, MacDonald D, Moloo H, Thavorn K, van Walraven C, Yang H, Forster AJ. Frailty as a Predictor of Death or New Disability After Surgery: A Prospective Cohort Study. Ann Surg. 2020 Feb;271(2):283-289. doi: 10.1097/SLA.0000000000002967. PMID 30048320
- [Background] Cameron ID, Fairhall N, Langron C, Lockwood K, Monaghan N, Aggar C, Sherrington C, Lord SR, Kurrle SE. A multifactorial interdisciplinary intervention reduces frailty in older people: randomized trial. BMC Med. 2013 Mar 11;11:65. doi: 10.1186/1741-7015-11-65. PMID 23497404
- [Background] de Labra C, Guimaraes-Pinheiro C, Maseda A, Lorenzo T, Millan-Calenti JC. Effects of physical exercise interventions in frail older adults: a systematic review of randomized controlled trials. BMC Geriatr. 2015 Dec 2;15:154. doi: 10.1186/s12877-015-0155-4. PMID 26626157
- [Background] Chan DC, Tsou HH, Yang RS, Tsauo JY, Chen CY, Hsiung CA, Kuo KN. A pilot randomized controlled trial to improve geriatric frailty. BMC Geriatr. 2012 Sep 25;12:58. doi: 10.1186/1471-2318-12-58. PMID 23009149